CLINICAL TRIAL: NCT03395119
Title: Efficacy of Fish Oil or Olive Oil Supplementation on the Health Effects of Ozone Exposure in Healthy Young Subjects
Acronym: OMEGOZ
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Environmental Protection Agency (EPA) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 15-2960
Record Dates: First submitted 2018-01-03; First posted 2018-01-10 (Actual); Last update posted 2021-01-15 (Actual); Status verified 2021-01

CONDITIONS: Healthy; Dietary Supplement
Keywords: Ozone exposure; Healthy Adults
MeSH Terms: interventions — Ozone; Fish Oils; Fatty Acids, Omega-3; Olive Oil

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Both participant and investigators are blinded for the assignment of dietary supplementation of fish oil, olive oil or control.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- No Supplements (Sham Comparator): The control group includes 20 healthy volunteers who will receive no supplements in the study. After 4 weeks, subjects will be exposed to clean air for 2 hours on the first day, then ozone for 2 hours on the second day
  Interventions: Drug: Ozone
- Fish oil (Experimental): Twenty healthy young adults will receive fish oil supplements for 4 weeks. After 4 weeks, subjects will be exposed to clean air for 2 hours on the first day, then ozone for 2 hours on the second day
  Interventions: Drug: Ozone; Dietary Supplement: Fish Oil
- Olive oil (Experimental): Twenty healthy young adults will receive olive oil supplements for 4 weeks. After 4 weeks, subjects will be exposed to clean air for 2 hours on the first day, then ozone for 2 hours on the second day
  Interventions: Drug: Ozone; Dietary Supplement: Olive Oil

INTERVENTIONS:
Drug: Ozone — After the four-week supplementation period, each subject will be blindly exposed on consecutive days to filtered air for 2 hours and to 0.3 ppm ozone for 2 hours, while undergoing intermittent moderate exercise (minute ventilation of 20 L/min/m²).
  Other Names: Filtered air
Dietary Supplement: Fish Oil — 3 (1-gram) soft-gels daily Commercially available, enteric-coated, soft-gels formulated to deliver >60% eicosapentaenoic/docosahexaenoic acids (EPA/DHA)
  Other Names: omega-3 fatty acids (eicosapentaenoic/docosahexaenoic)
  Arms: Fish oil
Dietary Supplement: Olive Oil — 3 soft-gels daily Commercially available soft-gels containing 1 gram of USDA organic certified, cold pressed, extra virgin, olive oil
  Other Names: extra virgin olive oil
  Arms: Olive oil

SUMMARY:
Purpose: A growing body of epidemiological data suggests an increased risk of cardiovascular events associated with air pollution. One of the common air pollutants, ozone, has been shown to induce oxidative stress and inflammation in the cardiovascular and respiratory systems. This proposed study is to examine the efficacy of fish oil and olive oil in modulating cardiovascular and pulmonary functions after ozone exposure. The objective is to understand the mechanistic basis for the health effects of ozone relative to those air pollutants. Treatment groups will include forty healthy young adults who will be given dietary supplementation of fish oil or olive oil. A control group will consist of 20 healthy volunteers who will receive no supplements. After 4 weeks, subjects will be exposed to clean air for 2 hours on the first day, then ozone for 2 hours on the second day. Cardiac rhythm, pulmonary function, vascular responses, endothelial function, and markers of coagulation and airway inflammation pre- and post- ozone exposure will be measured. This study is designed to build on the previous nutritional supplement interventional studies (UNC IRB # 07-0190 and UNC IRB # 11-1807), in order to understand the mechanism of action of particulate pollutants in comparison to that of ozone, a known oxidant air contaminant.

Participants: A total of sixty healthy 18-35 year-old male and female subjects will be involved in the study.

Procedures (methods): Forty healthy young adults will receive dietary supplementation consisting of fish oil or olive oil for 4 weeks. The control group includes 20 healthy volunteers who will receive no supplements in the study. After 4 weeks of supplementation or control regiment, each subject will be exposed to clean air for 2 hours on the first day, then ozone for 2 hours on the second day.

DETAILED DESCRIPTION:
Ozone pollution is a common problem across the world, including in the US. This proposed study is to examine the efficacy of fish oil and olive oil in modulating cardiovascular and pulmonary functions after ozone exposure. Results from this study will also increase our understanding of how ozone exposure adversely affects the functioning of the human cardiovascular and respiratory systems. This understanding may be especially important for patients with cardiopulmonary diseases.

Approximately 60 people will participate in this study.

You should expect to be in this study for about a month, but your participation could possibly last for 6 months. There are 4 sessions, including a consenting session (today) which will last for about 4 hours. The two exposure-day sessions will last approximately 8-9 hours each. There will also be an approximately 3-hour follow-up visit the day after your last exposure.

What will happen if you take part in the study? Before you agree to participate in this study, you must read the consent forms in their entirety. The research and medical staff will then answer all your questions and explain all the risks involved in this study to your satisfaction.

You should have already undergone a general physical examination to ensure that you are a suitable candidate for this study. If you are a female, you will be asked about your menstrual history. For all other female participants, a pregnancy test will be performed today, and this will be repeated on the exposure day if more than 7 days since last pregnancy test.

Consenting Day We will go over the study in detail so that you will know what we will expect from you as a participant and what you should expect from us as investigators. If you agree to participate in the study, you will sign all study consent forms and receive one set of signed copies.

You will have a breathing test (spirometry). You will breathe through a filter into a plastic device. Your lung function test results should meet certain criteria (Both Forced Vital Capacity (FVC) and Forced Expiatory Volume at the 1st second (FEV1) are equal to and greater than 80% of the reference value) to allow you to participate in the study.

You will undergo a procedure for for induced sputum. If you are a non-producer or the quality of the induced sputum sample that you produce does not meet the study criteria (we will know the sputum quality in the next two days), we will exclude you from the study. If that happens, you will be reimbursed for the time and procedures for the consenting session. If you qualify, you will be given instructions to prepare for the exposure sessions. Then you will be scheduled for the exposure sessions.

You will be give dietary supplementation of fish oil, olive oil or placebo for 4 weeks. Dietary and medication instructions will be given to restrict certain types of food and medicines during the supplementation period.

Exposure days We will call you a few days before the exposure session to remind you of your scheduled visit. You should avoid smoke, fumes, alcohol, and strenuous exercise 24 hours prior to all visits, and abstain from pan fried or grilled meat after midnight of the exposure day.

You will be asked to eat a light breakfast and arrive at the EPA medical station by 7:30 am. Please understand that it is very important that you arrive by this time in order for the study team to process all of the samples and data. Please note that we may have to cancel your participation if you arrive late.

Prior to exposure, you will:

* Have your vital signs checked (heart rate, respiratory rate, blood pressure, oxygen saturation level, and fill out a symptom questionnaire electronically).
* Have your heart rhythm recorded by a Holter monitor. You will have (10) electrocardiogram (ECG) leads attached to your chest. It may be necessary to clean and shave the areas of your chest where these leads will be placed. Excessive deodorant, skin lotions, and body sprays may interfere with the function of some of these leads. Therefore, we ask you to not apply these to your chest area on the day you report to the HSF. The leads will be connected to 2 monitors (small recording devices about the size and weight of a cell phone) to obtain readings of your heart rate and rhythm. It is preferable that the electrodes will stay in place for approximately 2 ½ days as you will have this measured several times during the study, however, you will be given the option to remove the electrodes by the end of each exposure day. You will be asked to recline quietly for 30 minutes while collecting your heart rhythm. It is important that you do not fall asleep during this 30-minute period. These measurements will allow us to determine whether wood smoke exposure causes small changes in the ability of your nervous system to regulate how your heart beats.
* Have the diameter of an artery in your upper arm measured by an ultrasound machine (BAU). The ultrasound operator will scan your arm with a probe and then place a tourniquet on your arm, much like a cuff used to measure blood pressure. Measurement of the size of the artery will be made two times. First, you will be asked to rest quietly for 15 minutes, and then the first 90 second scan will be performed. Then the blood pressure cuff on your arm will be inflated for 5 minutes in order to temporarily stop the flow of blood. You may feel sensations similar to that when your foot "goes to sleep", such as "pins and needles" and tingling. After the pressure cuff is released, a second scan will be taken of the artery.
* Have your retinas imaged using an ophthalmic camera before and after each exposure, and on the follow-up visit. You will be asked to place your chin on a rest in front of the camera. We will take pictures of the inside of both of your eyes. Glasses or contacts have to be removed for this test. Please bring your own contact lens container and solutions.
* Approximately 60 ml blood drawn (about 4 tablespoons) before and after each exposure, and on the follow-up visit. We will test this blood to see if wood smoke affects the ability of your blood cells to function. A small portion of the blood sample will be used to measure the relative content of various fatty acids present in your blood. With your permission, we also store some of the blood that we obtain during the study for yet-to-be-determined tests in the future.
* Have a breathing test (spirometry).
* Enter the exposure chamber and be exposed to filtered air or ozone.

During the exposure, you will:

• Undergo exposure for 2 hours to either clean filtered air or ozone in the chamber. You will receive clean filtered air on one day and ozone on the other day. You will not be given the information of the sequence of the exposure. Chamber conditions will be at a comfortable temperature and relative humidity. You will do mild exercise on a stationary bicycle in the chamber every other 15 minutes alternating with resting period for a total of 1 hour of exercise per chamber exposure. The target ventilation rate will be maintained at 20 L/min/ m2 and monitored by using pneumotach method. A study coordinator or other trained person will be seated outside the chamber observing you at all times. During the exposure, your heart will be monitored and the amount of oxygen present in your blood will be monitored by placing a device (pulse oximeter) on your finger. If it appears you are experiencing significant discomfort, breathing or heart problems, the exposure will be terminated immediately. In addition, you may elect to terminate the exposure at any time for any reason. If you do so, you will be paid in full for that day's session but will be ineligible for further participation in the study and any payments you would have received for future participation.

Immediately following the exposure, you will repeat the pre-exposure procedures and have a low fat lunch brought by you.

* Once you complete the above procedures, you will have about 1-2 hour waiting time before the next procedure. You can bring your personal laptop or books to use during that time. You will not be able to eat any food during this break time.
* Have samples of your airway secretions collected using the induced sputum procedure. You will be asked to breathe in different saline solutions (up to 5%) to help you expectorate. We will coach you on the procedure. First, you will gargle and clear your throat, and the cough up samples from deep in your chest and spit them into a cup. Your lung function will be monitored during the procedure. Food must be avoided for 2 hours prior to this test.
* Be assessed and discharged by the study personnel.

Follow up visit (about 3 hours) You will return to the HSF the next morning (approximately 18 hours after your 2nd exposure) and you will repeat the pre-exposure procedures.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-35 years old healthy male and female (19≤BMI≤30).
* Physical conditioning allowing intermittent, moderate exercise for 2 hours, and ability to complete the exposure exercise regimen chosen to induce a minute ventilation rate of 20 L/min/m² for 15 minutes without exceeding 80% of predicted maximal heart rate.
* Normal resting electrocardiography (ECG)
* Normal lung function
* Oxygen saturation greater than 94% at the time of physical exam.
* Individuals whose blood omega-3 index is 5% or lower at the time of screening.

Exclusion Criteria:

1. Individuals with a history of acute or chronic cardiovascular disease, chronic respiratory disease, cancer (possible exception for history of non-melanoma skin cancer), rheumatologic disease, neuromuscular disease, or immunodeficiency state.
2. Individuals with a cardiovascular disease risk score greater than 10% using the American College of Cardiology and the American Heart Association Atherosclerotic Cardiovascular Disease risk calculator. (Based on the 10-year risk of heart disease or stroke using the Atherosclerotic Cardiovascular Disease algorithm published in 2013 American College of Cardiology/American Heart Association Guideline on the Assessment of Cardiovascular risk.)
3. Uncontrolled hypertension (>150 systolic, >90 diastolic).
4. Individuals who are diabetic (previously diagnosed or with hemoglobin A1c level >6.4%).
5. Individuals with asthma or a history of asthma.
6. Individuals who are allergic to chemical vapors or gases.
7. Individuals who have skin allergy to tape or electrodes.
8. Individuals is pregnant, attempting to become pregnant or breastfeeding.
9. Individuals who are currently smoking (including vaping, hookah and e-cigarette) or have smoking history within 1 year of study (defined as more than 1 pk/yr in the past year) or have a greater than/equal to a 5 pack year smoking history.
10. Individuals living with a smoker who smokes inside the house.
11. Individuals who are regularly exposed to high levels of vapors, dust, gases, or fumes.
12. Individuals that do not understand or speak English.
13. Individuals that are unable to perform the exercise required for the study.
14. Individuals who are taking Î2-blocker medications.
15. Individuals who are allergic to fish or omega-3 fatty acids, or are on prescription of taking omega-3 fish oil as therapy.
16. Individuals that are unwilling or unable to stop taking medications that may impact the results of ozone challenge for the duration of the study. Medications not specifically mentioned here may be reviewed by the investigators prior to an individuals inclusion in the study.
17. Individuals who are unwilling or unable to stop taking any current dietary supplements for the duration of the study. Prebiotics and probiotics are acceptable.
18. Individuals who are unwilling or unable to adhere to study specific dietary restrictions (see details under A.4.2 dietary instruction).
19. Individuals who have unspecified illnesses, which in the judgment of the investigators might increase the risk associated with ozone inhalation will be a basis for exclusion.
20. Individuals with bleeding/clotting disorders.
21. Individuals who are not willing to participate the induced sputum procedure on the training day.

Temporary exclusion criteria:

1. Individuals who have recent (within 6 month) abdominal and/or eye surgery, or with any types of hernia, as well as any other contraindications for raised intra-abdominal pressure.
2. Individuals who have had an acute respiratory illness within 4 weeks.
3. Individuals who are currently taking systemic steroids, oral anticoagulants, over-the counter pain medications (such as aspirin, Advil, Aleve) or nonsteroidal anti-inflammatory drugs, or have taken these medications within the last 14 days.
4. Individuals who have active allergies.

Use of other medications will be evaluated on a case-by-case basis. There is the potential that an individuals current medication use will preclude them from participating in the study at the current time, but they may be reassessed and potentially rescheduled for participation at a later time.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2017-12-18 (Actual); Primary Completion 2020-12-18 (Actual); Study Completion 2020-12-18 (Actual)

PRIMARY OUTCOMES:
Change in forced expired volume in the first second (FEV1) from air exposure (Day 1) to ozone exposure (Day 2) | Day 1, Day 2
  FEV1 is determined by spirometry

SECONDARY OUTCOMES:
endothelial cell function 1 hour post-exposure | 1 hour pre-exposure, 1 hour post-exposure
  Brachial artery ultrasound will be used to evaluate flow-mediated dilatation which will be performed in the Human Studies Facility (HSF) at U.S. Environmental Protection Agency (EPA) using an ultrasound instrument. The diameter of the brachial artery will be measured at baseline and during reactive hyperemia.
endothelial cell function 18 hour post-exposure | 1 hour pre-exposure, 18 hour post-exposure
  Brachial artery ultrasound will be used to evaluate flow-mediated dilatation which will be performed in the HSF at EPA using an ultrasound instrument. The diameter of the brachial artery will be measured at baseline and during reactive hyperemia.
diameters of retinal arteries and veins 1 hour post-exposure | 30 min pre-exposure, 1 hour post-exposure
  Retinal images will be taken using an FDA-approved, commercially available, non-mydriatic fundus camera. Images will be taken from both eyes.
diameters of retinal arteries and veins 18 hour post-exposure | 30 min pre-exposure, 18 hour post-exposure
  Retinal images will be taken using an FDA-approved, commercially available, non-mydriatic fundus camera. Images will be taken from both eyes.
airway inflammation 4 hour post-exposure | 6 weeks prior to the exposure, 4 hour post-exposure
  Sputum induction will be performed to determine the airway inflammation.
Heart rate variability 1 hour post-exposure | 1 hour pre-exposure, 1 hour post-exposure
  Heart rate variability will be collected by the Holter monitor.
Heart rate variability 18 hour post-exposure | 1 hour pre-exposure, 18 hour post-exposure
  Heart rate variability will be collected by the Holter monitor.
Blood fatty acids 2 hour post-exposure | 6 weeks prior to the exposure, 2 hours pre-exposure
  Blood sample will be collected for fatty acids analysis
Blood fatty acids 30 min post-exposure | 2 hour pre-exposure, 30 min post-exposure
  Blood sample will be collected for fatty acids analysis
Blood fatty acids 18 hour post-exposure | 2-hour pre-exposure, 18 hour post-exposure
  Blood sample will be collected for fatty acids analysis
Blood cholesterol 2 hour post-exposure | 6 weeks prior to the exposure, 2 hours pre-exposure
  Blood sample will be collected for measuring the cholesterol level
Blood cholesterol 30 min post-exposure | 2 hour pre-exposure, 30 min post-exposure
  Blood sample will be collected for measuring the cholesterol level
Blood cholesterol 18 hour post-exposure | 2-hour pre-exposure, 18 hour post-exposure
  Blood sample will be collected for measuring the cholesterol level
Forced expired volume in the first second (FEV1) 18 hour post-exposure | immediate post-exposure to ozone within 30 min, 18 hour post-exposure
  Forced expired volume in the first second (FEV1) is determined by the spirometry

CONTACTS AND LOCATIONS:
Overall Officials: James Samet, PhD, Principal Investigator — Environmental Protection Agency, University of North Carolina at Chapel Hil
Locations (1):
- U.S. Environmental Protection Agency Human Studies Facility, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data will be shared through the U.S. EPA's ScienceHub database. ScienceHub is used to upload and store datasets associated with journal articles. Non-sensitive datasets are then made publicly accessible via the Environmental Dataset Gateway in fulfillment of the EPA's requirement to adhere to the Office of Management and Budget's Open Data Policy.
Time Frame: Data will be available in ScienceHub after the publication of the study is completed.
Access Criteria: Data will be available to the public